CLINICAL TRIAL: NCT01031199
Title: Open-label, Non-randomized, Positron Emission Tomography (PET) Imaging Study to Evaluate a Single Dose of 140 MBq (ca. 5 mSv) ZK 6032924 (BAY85-8101) for Its Diagnostic Potential in Either Drug-naïve or Specifically (IFN-beta) Pretreated Patients With Multiple Sclerosis (MS) With Acute Relapse or Patients With Clinically Isolated Syndrome (CIS), Compared to Healthy Volunteers
Brief Title: Evaluation of the Positron Emission Tomography (PET) Tracer ZK 6032924 in Patients With Multiple Sclerosis Compared to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 13101; 2008-000981-22 (EudraCT Number)
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-04

CONDITIONS: Positron-Emission Tomography; Multiple Sclerosis
Keywords: Multiple sclerosis; Diagnostic imaging; Neuroinflammation; PET diagnosis; PET tracer
MeSH Terms: conditions — Multiple Sclerosis; Neuroinflammatory Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: F-18 FEDAA1106 (BAY85-8101)
- Arm 2 (Experimental)
  Interventions: Drug: F-18 FEDAA1106 (BAY85-8101)

INTERVENTIONS:
Drug: F-18 FEDAA1106 (BAY85-8101) — MS/CIS patients: Single intravenous bolus of 140 MBq BAY85-8101 ± 15% (ca. 5 mSv), applied mass of tracer < 5 µg, PET
  Arms: Arm 1
Drug: F-18 FEDAA1106 (BAY85-8101) — Healthy controls: Single intravenous bolus of 140 MBq BAY85-8101 ± 15% (ca. 5 mSv), applied mass of tracer < 5 µg, PET
  Arms: Arm 2

SUMMARY:
PET (positron emission tomography) imaging with BAY85-8101 for investigation in patients with Multiple Sclerosis compared to healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers for brain imaging:

* males or females, age 20 - 55 years
* assessment of the brain MRI as "normal (age-appropriate)"
* absence of any sign of CNS disease, no co-medi cation Patients for brain imaging
* males or females, age 20 - 55 years
* patients with previously diagnosed MS, presenting with acute relapse, without any current immunomodulating therapy for MS ("drug-naïve"), or patients presenting with first clinical episode suggestive of demyelinating disease (Clinically Isolated Syndrome, CIS)
* patients with previously diagnosed MS, presenting with acute relapse, receiving currently immunomodulatory therapy exclusively with interferon β
* MRI: >/= 2 T2 lesions and >/= 1 Gadolinium- (Gd-) enhancing lesion

Exclusion Criteria:

Exclusion criteria for all healthy volunteers and patients:

* Pregnancy or lactation
* Any disease, condition, or concomitant medications that significantly compromises the function of the body systems and could result in excessive accumulation, impaired metabolism, altered excretion of the radiotracer, or might interfere with the conduct of the study or interpretation of the results
* other forms of diseases with neuroinflammatory components

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Standard quantification variables derived from 3D PET imaging and brain modeling. | Day of study tracer administration
Visual analysis/description of the uptake and description of brain PET scans. | Day of study tracer administration

SECONDARY OUTCOMES:
Standard Safety Parameter: Adverse Event Collection | maximum time from Screening to Follow-up are 37days
Standard Safety Parameter: Electrocardiogram | maximum time from Screening to Follow-up are 37days
Standard Safety Parameter: Safety laboratory | maximum time from Screening to Follow-up are 37days
Standard Safety Parameter: Vital signs | maximum time from Screening to Follow-up are 37days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Heidelberg, Victoria, Australia
- Stockholm, Sweden

REFERENCES:
- [Derived] Takano A, Piehl F, Hillert J, Varrone A, Nag S, Gulyas B, Stenkrona P, Villemagne VL, Rowe CC, Macdonell R, Tawil NA, Kucinski T, Zimmermann T, Schultze-Mosgau M, Thiele A, Hoffmann A, Halldin C. In vivo TSPO imaging in patients with multiple sclerosis: a brain PET study with [18F]FEDAA1106. EJNMMI Res. 2013 Apr 24;3(1):30. doi: 10.1186/2191-219X-3-30. PMID 23618062